CLINICAL TRIAL: NCT03360760
Title: Presurgical Chemotherapy Compared With Immediate Surgery and Adjuvant Chemotherapy for Nonmetastatic Osteosarcoma of the Pelvis and Sacrum
Brief Title: Timing of Surgery in Nonmetastatic Osteosarcoma of the Pelvis and Sacrum
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, GUO WEI, Director of Musculoskeletal Tumor Center, Peking University People's Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PKUPH-sarcoma 04
Record Dates: First submitted 2017-11-26; First posted 2017-12-04 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Osteosarcoma of Pelvis
Keywords: osteosarcoma; pelvis; sacrum
MeSH Terms: conditions — Osteosarcoma | interventions — Doxorubicin; Cisplatin; Methotrexate; Ifosfamide; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre surgical Chemotherapy (Experimental): Immediate pre surgical chemotherapy treated with four drugs including doxorubicin, cisplatin, high-dose methotrexate (MTX) and ifosfamide in eleven weeks, and then definitive surgery followed by adjuvant chemotherapy according to chemotherapy regimen in Peking University People's Hospital(PKUPH).
  Interventions: Drug: Doxorubicin; Drug: Cisplatin; Drug: Methotrexate; Drug: Ifosfamide; Procedure: definitive surgery; Other: pre surgical chemotherapy
- Immediate Surgery (Other): Immediate definitive surgery, and then post operative chemotherapy based on doxorubicin, cisplatin, high-dose MTX and ifosfamide according to chemotherapy regimen in PKUPH.
  Interventions: Drug: Doxorubicin; Drug: Cisplatin; Drug: Methotrexate; Drug: Ifosfamide; Procedure: definitive surgery

INTERVENTIONS:
Drug: Doxorubicin — 60mg/m^2, in the adjuvant chemotherapy regimen for osteosarcoma in PKUPH
  Other Names: Adriamycin
Drug: Cisplatin — 100mg/m^2, in the adjuvant chemotherapy regimen for osteosarcoma in PKUPH
  Other Names: cisplatinum; platamin
Drug: Methotrexate — High dose of methotrexate (8-12g/m^2), in the adjuvant chemotherapy regimen for osteosarcoma in PKUPH
  Other Names: HD-MTX
Drug: Ifosfamide — 12g/m^2, in the adjuvant chemotherapy regimen for osteosarcoma in PKUPH
  Other Names: ifosphamide
Procedure: definitive surgery — Including limb-sparing procedure and amputation
Other: pre surgical chemotherapy — chemotherapy that given before definitive surgery
  Other Names: neoadjuvant chemotherapy
  Arms: Pre surgical Chemotherapy

SUMMARY:
To study the effect of the timing of surgery on outcome of patients with nonmetastatic osteosarcoma of pelvis and sacrum.

DETAILED DESCRIPTION:
Successful therapeutic interventions to prevent disease progression in patients with nonmetastatic osteosarcoma of pelvis and sacrum have included surgery with adjuvant chemotherapy. Pre-surgical chemotherapy has been advocated for these patients because of putative improvement in event-free survival (EFS). The advantages of pre-surgical chemotherapy include early administration of systemic chemotherapy, shrinkage of primary tumor, and pathologic identification of risk groups. The theoretic disadvantage is that it exposes a large tumor burden to marginally effective chemotherapy, especially in the axial region. The contribution of chemotherapy and surgery timing has not been tested rigorously. To study the effect of the timing of surgery on outcome of patients with nonmetastatic osteosarcoma of pelvis and sacrum, we conducted multicenter randomized trial to determine whether chemotherapy administered before definitive resection of primary tumors improved EFS and overall survival compared with traditional resection of the primary tumor followed by adjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age >10 years and <40 years;
* High-grade nonmetastatic osteosarcoma in pelvis or sacrum;
* Diagnosis confirmed histologically and reviewed centrally;
* No evidence of metastatic disease with computed tomography scan of the chest and radionuclide bone scan, or Positron Emission Tomography (PET/CT) within 2 weeks of entry;
* No prior therapy;
* Eastern Cooperative Oncology Group performance status 0-1;
* Life expectancy >3 months;
* Adequate renal, hepatic, and hemopoietic function;

Exclusion Criteria:

* Previously treated by chemotherapy or unplanned surgery in other hospital;
* Have had other kinds of malignant tumors at the same time;
* Uncontrolled complications, such as diabetes mellitus and so on;
* Intravascular tumor thrombus on enhanced CT or magnetic resonance (MR);
* Unresectable disease evaluated by surgeons.

Ages: 10 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | 5 years
  Calculated from the date of treatment start until death, whichever comes first.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 5 years
  Calculated from the date of treatment start until the time of disease progression or death, whichever comes first.
Tumor necrosis rate | 5 years
  The percentage of tumor necrosis calculated in the resected specimen in Arm 2.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Guo, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Undecided